CLINICAL TRIAL: NCT00599196
Title: An Open-Label Extension to the Double-Blind SP513 Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Subjects With Early-Stage Idiopathic Parkinson's Disease
Brief Title: An Open-Label Extension Trial to Assess the Safety of Long-Term Treatment of Rotigotine in Early-Stage Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0716; SP513OL (Other: UCB)
Record Dates: First submitted 2007-12-24; First posted 2008-01-23 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2010-09

CONDITIONS: Early Stage Parkinson's Disease
Keywords: Rotigotine; Neupro®
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): Rotigotine
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine trans-dermal patches, once daily:
  10 cm2 (2 mg/24 hours); 20 cm2 (4 mg/24 hours); 30 cm2 (6 mg/24 hours); 40 cm2 (8 mg/24 hours); 50 cm2 (10 mg/24 hours); 60 cm2 (12 mg/24 hours); 70 cm2 (14 mg/24 hours); 80 cm2 (16 mg/24 hours);
  Optimal dosing:
  During the first year: The maximum Rotigotine dose allowed is 8 mg/24 hours.
  After the first year: allowed dose increase of rotigotine up to a maximum of 16 mg/24 hours.
  Other Names: Neupro®

SUMMARY:
The objective of this open-label extension is to assess the safety and tolerability of long-term treatment of the rotigotine patch in subjects with early-stage idiopathic Parkinson's disease

DETAILED DESCRIPTION:
This is the open-label extension to the randomized, double-blind, placebo- and ropinirole-controlled SP513 trial that assessed the efficacy and safety and tolerability of the Rotigotine patch in subjects with early-stage idiopathic Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed six months of maintenance treatment in the SP513 double-blind trial

Exclusion Criteria:

* Subjects who had an ongoing serious adverse event from SP513 double-blind trial that was assessed as related to study medication

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2002-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (63):
- Australia (4):
  - Concord
  - Darlinghurst
  - East Gosford
  - Westmead
- Austria (2):
  - Innsbruck
  - Vienna
- Belgium (2):
  - Brussels
  - Hoboken
- Zagreb, Croatia
- Czechia (3):
  - Brno
  - Ostrava
  - Pilsen
- Finland (5):
  - Espoo
  - Kuopio
  - Lappeenranta
  - Oulu
  - Pori
- France (3):
  - Aix-en-Provence
  - Caen
  - Toulouse
- Germany (4):
  - Aachen
  - Dresden
  - Kiel
  - Marburg
- Hungary (3):
  - Budapest
  - Miskolc
  - Pécs
- Israel (3):
  - Hadera
  - Petah Tikva
  - Tel Aviv
- Italy (3):
  - Milan
  - Padua
  - Pozzilli
- Netherlands (2):
  - Breda
  - Geldrop
- New Zealand (4):
  - Auckland
  - Christchurch
  - North Shore
  - Wellington
- Norway (2):
  - Stavanger
  - Trondheim
- Poland (7):
  - Gdansk
  - Katowice
  - Krakόw
  - Lublin
  - Mosina k/Poznania
  - Olsztyn
  - Warsaw
- South Africa (2):
  - Cape Town
  - Pretoria
- Spain (2):
  - Barcelona
  - Pamplona
- Sweden (2):
  - Karlstad
  - Stockholm
- Switzerland (2):
  - Bern
  - Lausanne
- United Kingdom (7):
  - Birmingham
  - Blackpool
  - Glasgow
  - Liverpool
  - London
  - Newcastle upon Tyne
  - Swansea

REFERENCES:
- [Derived] Giladi N, Boroojerdi B, Surmann E. The safety and tolerability of rotigotine transdermal system over a 6-year period in patients with early-stage Parkinson's disease. J Neural Transm (Vienna). 2013 Sep;120(9):1321-9. doi: 10.1007/s00702-013-1001-5. Epub 2013 Mar 19. PMID 23508526
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An Open-Label Extension to Assess the Safety of Long-Term Treatment of Rotigotine in Subjects with Early-Stage Idiopathic Parkinson's Disease from August 2002 to December 2008
Pre-assignment Details: One subject was excluded from the safety set because he withdrew consent prior to receiving any Open Label study medication.
Groups:
- Rotigotine: Optimal dosing for Rotigotine transdermal patches, once daily: Year 1, the maximum dose allowed is 8 mg/24 hours. After Year 1, a dose increase is allowed up to a maximum of 16 mg/24 hours.
Period: Overall Study
Arm/Group | Rotigotine
Started | 381
Completed | 0 (Study fully recruited. Completed upon market authorization and commercial availability of Neupro.)
Not Completed | 381
Not completed — Lack of Efficacy | 22
Not completed — Adverse Event | 93
Not completed — Unsatisfactory compliance of subject | 3
Not completed — Subject withdrew consent | 43
Not completed — Study ended per sponsor | 197
Not completed — Lost to Follow-up | 17
Not completed — Other: Patient Leaving For Israel | 1
Not completed — Other: Spouse Withdrew Consent | 1
Not completed — Other: Diagnosis No Longer Idiopathic Pd | 1
Not completed — Other: Pt Moved To Australia | 1
Not completed — Other: Patient Stopped Due To Moving | 1
Not completed — Other: Inv Switched Dopamine Agonist | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rotigotine
Number analyzed (Participants) | 380
Age, Categorical [Count of Participants; unit: Participants] — Of the 381 subjects who entered the study, 380 are included in this summary based on the Safety Set (SS). One subject was excluded from the Safety Set because he withdrew consent prior to receiving any Open Label study medication.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 215
    >=65 years | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 230
Region of Enrollment [Number; unit: participants]
  Finland | 16
  Spain | 10
  Austria | 12
  Israel | 30
  United Kingdom | 38
  Italy | 9
  Switzerland | 4
  France | 10
  Czech Republic | 44
  Hungary | 17
  Poland | 65
  Belgium | 12
  Croatia | 17
  Australia | 7
  South Africa | 42
  Germany | 7
  Norway | 4
  Netherlands | 5
  New Zealand | 19
  Sweden | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event During This Open-label Extension Study
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: six years
Population: Of the 381 subjects who entered the study, 380 are included in this summary based on the Safety Set (SS). One subject was excluded from the safety set because he withdrew consent prior to receiving any Open Label study medication.
Measure: Number; unit: Subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 380
Subjects | 369

2. Secondary Outcome: Number of Subjects Who Withdrew From the Trial Due to an Adverse Event
Description: as for outcome 1
Time Frame: six years
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Rotigotine
Number analyzed (Participants) | 380
Subjects | 93

3. Secondary Outcome: Mean Epworth Sleepiness Scale Score During the Open-label Extension
Description: The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. The total ESS score is the sum of 8 item-scores and can range between 0 and 24. The higher the score, the higher the person's level of daytime sleepiness.
Time Frame: Visit 10 (end of year 1), Visit 14 (end of year 2), Visit 18 (end of year 3), Visit 22 (end of year 4), Visit 26 (end of year 5), Visit 30 (end of year 6), End of Treatment (last study visit or early withdrawal visit)
Population: Of the 380 subjects who are included in the Safety Set (SS), 5 subjects discontinued prior to entering the maintenance phase (n=375), however 2 of these subjects returned for the End of Treatment visit (n=377). Last observation carried forward (LOCF) was utilized for subjects who entered the maintenance phase.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Rotigotine
Number analyzed (Participants) | 377
Score on a scale
  Visit 10 (end of year 1) (n=375) | 5.8 (3.8)
  Visit 14 (end of year 2) (n=375) | 6.2 (4.1)
  Visit 18 (end of year 3) (n=375) | 6.7 (4.5)
  Visit 22 (end of year 4) (n=375) | 6.7 (4.6)
  Visit 26 (end of year 5) (n=375) | 6.7 (4.5)
  Visit 30 (end of year 6) (n=375) | 6.8 (4.5)
  End of Treatment (n=377) | 6.8 (4.5)

ADVERSE EVENTS:
Time Frame: up to 6 years
Arm/Group | Rotigotine
Serious Adverse Events (participants affected / at risk) | 131/380
Other Adverse Events (participants affected / at risk) | 323/380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=380)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 10 (11)
Angina pectoris (Cardiac disorders) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Application site irritation (General disorders) | 1 (1)
Application site rash (General disorders) | 1 (1)
Application site erythema (General disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
Hernia (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Therapeutic response decreased (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 5 (5)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 2 (2)
Hepatic cyst (Hepatobiliary disorders) | 1 (1)
Biliary tract disorder (Hepatobiliary disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Bronchitis acute (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Appendicitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (3)
Influenza (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (3)
Viral infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 9 (13)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 6 (7)
Femur fracture (Injury, poisoning and procedural complications) | 5 (5)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Skin injury (Injury, poisoning and procedural complications) | 1 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 (12)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Toe deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parkinson's disease (Nervous system disorders) | 9 (10)
Somnolence (Nervous system disorders) | 1 (1)
Syncope vasovagal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Sudden onset of sleep (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Movement disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Myelitis transverse (Nervous system disorders) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 4 (4)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Sleep attacks (Psychiatric disorders) | 2 (3)
Paranoia (Psychiatric disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2)
Impulse-control disorder (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 2 (3)
Ankle operation (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Cataract operation (Surgical and medical procedures) | 2 (2)
Cholecystectomy (Surgical and medical procedures) | 2 (2)
Colostomy closure (Surgical and medical procedures) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1)
Deep brain stimulation (Surgical and medical procedures) | 1 (1)
Lung lobectomy (Surgical and medical procedures) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1)
Cardiovascular insufficiency (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Thrombophlebitis (Vascular disorders) | 1 (1)
Aortic aneurysm (Vascular disorders) | 2 (2)
Femoral arterial stenosis (Vascular disorders) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=380)
Nausea (Gastrointestinal disorders) | 72 (115)
Vomiting (Gastrointestinal disorders) | 25 (30)
Constipation (Gastrointestinal disorders) | 34 (36)
Diarrhoea (Gastrointestinal disorders) | 20 (21)
Application site reaction (General disorders) | 45 (54)
Application site pruritus (General disorders) | 27 (32)
Application site erythema (General disorders) | 26 (27)
Oedema peripheral (General disorders) | 71 (93)
Fatigue (General disorders) | 26 (30)
Urinary tract infection (Infections and infestations) | 29 (41)
Nasopharyngitis (Infections and infestations) | 24 (33)
Influenza (Infections and infestations) | 20 (22)
Fall (Injury, poisoning and procedural complications) | 43 (81)
Weight increased (Investigations) | 19 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 57 (78)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 (48)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 (21)
Somnolence (Nervous system disorders) | 146 (234)
Dizziness (Nervous system disorders) | 51 (62)
Headache (Nervous system disorders) | 29 (32)
Parkinson's disease (Nervous system disorders) | 23 (35)
Insomnia (Psychiatric disorders) | 48 (57)
Depression (Psychiatric disorders) | 38 (45)
Hallucination (Psychiatric disorders) | 21 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (31)
Hypertension (Vascular disorders) | 41 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.